CLINICAL TRIAL: NCT00672997
Title: A Six-Week, Multi-Center, Double-Masked, Safety and Efficacy Study of Travoprost 0.004%/Timolol 0.5% BAC-free Compared to Travoprost 0.004%/Timolol 0.5% in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Phase III Study of Travoprost/Timolol Combination in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-64
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — Travoprost; Timolol; Ophthalmic Solutions; Duotrav

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost/Timolol BAC-free (Experimental): Travoprost 0.004%/Timolol 0.5% BAC-free ophthalmic solution, 1 drop in each eye, once daily (QD) at 9 AM (±30 minutes), for 6 weeks
  Interventions: Drug: Travoprost 0.004%/Timolol 0.5% BAC-free ophthalmic solution
- Travoprost/Timolol (Active Comparator): Travoprost 0.004%/Timolol 0.5% ophthalmic solution, 1 drop in each eye, once daily (QD) at 9 AM (±30 minutes), for 6 weeks
  Interventions: Drug: Travoprost 0.004%/Timolol 0.5% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004%/Timolol 0.5% BAC-free ophthalmic solution
  Arms: Travoprost/Timolol BAC-free
Drug: Travoprost 0.004%/Timolol 0.5% ophthalmic solution
  Other Names: DuoTrav®
  Arms: Travoprost/Timolol

SUMMARY:
The purpose of this study is to demonstrate equivalent safety and IOP-lowering effectiveness of two Travoprost/Timolol combination products in patients diagnosed with open-angle glaucoma or ocular hypertension. This global study will be conducted in the US (C-07-64, NCT00672997) and Japan (C-08-08, NCT00760539).

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma or confirmed ocular hypertension.
* Mean IOP in at least one eye, the same eye(s):22-36 mmHg at 9 AM on eligibility visits 1 & 2 and 21-36 mmHg at 11 AM and 4 PM on Eligibility Visits 1 & 2.
* Sign an informed consent form.
* Discontinued use of all IOP-lowering medications(s) for a minimum of 4 days to a minimum of 27 days or more prior to the Eligibility 1 Visit.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, planning to become pregnant during the study period, breast-feeding, or not using adequate birth control measures.
* Any form of glaucoma other than open-angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component) or confirmed ocular hypertension.
* History or current evidence of chronic or recurrent severe inflammatory eye disease in either eye.
* History or current evidence of clinically relevant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment in either eye.
* Best-corrected visual acuity (BCVA) worse than 0.6 logMAR in either eye.
* Severe central visual field loss in either eye.
* Not able to safely discontinue use of all IOP-lowering ocular medication(s) according to the Ocular Hypotensive Medication Washout Schedule.
* History or current evidence of bronchial asthma, or severe chronic obstructive pulmonary disease (COPD) that would in the opinion of the investigator preclude the safe administration of a topical beta-blocker.
* History or other evidence of severe illness or any other conditions which would make the subject, in the opinion of the investigator, unsuitable for the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) combined across all visits and timepoints | Week 2 (9 AM, 11 AM, and 4 PM); Week 6 (9 AM, 11 AM, and 4 PM)
  IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Percentage of patients with IOP <18 mmHg or IOP percent reduction of ≥ 30% by visit | Week 2 (9 AM, 11 AM, and 4 PM); Week 6 (9 AM, 11 AM, and 4 PM)
  IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Smith, B.S., Study Director — Alcon Research